CLINICAL TRIAL: NCT04195100
Title: Local Application of Pilocarpine for Relieving Dry Mouth Complaints: A Randomized Controlled Pilot Trial
Brief Title: Local Pilocarpine for Relieving Dry Mouth
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: METC18-071
Record Dates: First submitted 2019-12-04; First posted 2019-12-11 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Patients of Advanced Age (≥ 70 Years) With a Clinical Diagnosis of Chronic Dry Mouth
Keywords: Xerostomia; Pilocarpine; advanced age (≥ 70 years)
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose pilocarpine (Active Comparator): low dose pilocarpine = 3 x 2.0 mg = 3 x 2 drops of pilocarpine 20.0 mg/ml (2%) per day
  Interventions: Drug: Pilocarpine Ophthalmic Solution
- High dose pilocarpine (Active Comparator): high dose pilocarpine = 3 x 5.0 mg = 3 x 5 drops of pilocarpine 20.0 mg/ml (2%) per day
  Interventions: Drug: Pilocarpine Ophthalmic Solution

INTERVENTIONS:
Drug: Pilocarpine Ophthalmic Solution — 1. low dose pilocarpine = 3 x 2.0 mg = 3 x 2 drops of pilocarpine 20.0 mg/ml (2%) per day
  2. high dose pilocarpine = 3 x 5.0 mg = 3 x 5 drops of pilocarpine 20.0 mg/ml (2%) per day

SUMMARY:
The investigators intended for this study to deliver the "proof-of-concept" that locally administered pilocarpine drops in two doses are effective in a population of elderly (aged ≥ 70 years) with xerostomia at the expense of limited adverse events. To this end, the study aims to quantify the effect size of pilocarpine in two different dosages. In case the investigators observe clinically meaningful changes in xerostomia through measured NRS, a sufficiently-powered RCT will be prepared to compare pilocarpine to placebo.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years of age
* Clinical diagnosis of chronic dry mouth defined as a Numeric Rating Scale (NRS) score ≥ 5 (scale 0 - 10, with 0 = no dry mouth and 10= worst possible dry mouth) on severity of xerostomia for more than 3 months.

Exclusion Criteria:

* Existence of cognitive impairment and/or diagnosis of dementia appraised by treating physician
* Inability to fill out the questionnaires due to other reasons
* Prior radiation therapy of the head-and-neck region
* Known m. Sjögren disease
* Contra-indications for parasympathicomimetics (uncontrolled asthma, acute heart failure, active peptic ulceration, known hypersensitivity to pilocarpine, and when miosis is undesirable, e.g., in acute iritis and in narrow-angle (angle closure) glaucoma.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in xerostomia score (Numeric Rating Scale) | 3 weeks
  The Numeric Rating Scale is used to quantify the level of severity of xerostomia using a 0-10 cm Numeric Rating Scale ranging from 0 = no dry mouth to 10 = worst possible dry mouth
Change in oral health-related quality of life (Dutch Geriatric Oral Health Assessment Index) | 2 weeks
  Questionnaires assessing Oral health-related quality of life of adults, in particular older people is measured 4 times during this study by the doctor/research nurse . It comprises 12 items that measure three dimensions of Oral health-related quality of life: physical function items, psychosocial function and pain/discomfort.

SECONDARY OUTCOMES:
Adverse effects | 3 weeks
  adverse events or other symptoms
Global perceived effect | 3 weeks
  The Global perceived effect scale asks the patient to rate, on a numerical scale, how much their condition has improved or deteriorated since some predefined time point.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke van den Beuken, Prof, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04195100/Prot_000.pdf